CLINICAL TRIAL: NCT05537675
Title: Semi-automated Segmentation Methods of SSTR PET for Dosimetry Prediction in Refractory Meningiomas Treated by SSTR-targeted Peptide Receptor Radionuclide Therapy
Brief Title: Semi-automated Segmentation Methods of SSTR PET for Dosimetry Prediction
Acronym: 177Lumen
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Antoine VERGER, Principal investigator, Central Hospital, Nancy, France
Other Study IDs: 2022PI
Record Dates: First submitted 2022-09-08; First posted 2022-09-13 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Refractory Meningioma
MeSH Terms: conditions — Meningioma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 20 patients with meningioma: 20 meningioma patients will be included in this study, 10 of whom will have been treated with Lutathera®.
  Interventions: Other: To evaluate the SUVmean (Standard Uptake Value) as a predictive factor of the tumor absorbed dose compared to the SUVmax
- 10 patients will have been treated with Lutathera®.: 10 patients of the 20 will have been treated with Lutathera®.
  Interventions: Other: To evaluate the SUVmean (Standard Uptake Value) as a predictive factor of the tumor absorbed dose compared to the SUVmax

INTERVENTIONS:
Other: To evaluate the SUVmean (Standard Uptake Value) as a predictive factor of the tumor absorbed dose compared to the SUVmax — Measure SUVmean (Standard Uptake Value) and SUVmax on PET exams

SUMMARY:
Tumor dosimetry with somatostatin receptor-targeted peptide receptor radionuclide therapy (SSTR-targeted PRRT) by 177Lutetium-DOTATATE might contribute to improve follow-up and treatment response of refractory meningiomas. This study aims to evaluate Standard Uptake Value mean (SUVmean) as a tumoral absorbed dose predictive predictive factor and propose semi-automated segmentation method to determine metabolic tumor volume with pretherapeutic 68-Gallium-DOTATOC PET.

ELIGIBILITY:
Inclusion Criteria:

* Patients with meningioma

Exclusion Criteria:

- PET scan not available

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 20 patients with meningioma will be included in this study, and 10 patients of 20 will have been treated with Lutathera®.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2022-11-06 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
To evaluate the SUVmean (Standard Uptake Value)as a predictive factor of the tumor absorbed dose compared to the SUVmax | 2 months
  Measurements of SUVmean and SUVmax at the lesion level on 68Ga-DOTATOC PET/CT Correlation between SUVmean and max measurements with tumor absorbed doses.
To propose a semi-automated segmentation | 1 month
  Propose a semi-automated segmentation method for determining metabolic tumor volume with pretherapy DOTATOC labelled with gallium-68 PET. (68Ga-DOTATOC PET)

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Sophie HUE, MSc, Study Director — CHRU Nancy
Locations (1):
- Nuclear medicine Department CHRU de NANCY, Vandœuvre-lès-Nancy, France